CLINICAL TRIAL: NCT02528968
Title: UK-PK Study: National Study of the Implementation of a Pharmacokinetic-Focused Educational Package for Patients Living With Severe Haemophilia A
Brief Title: National Study of a Pharmacokinetic-Focused Educational Package for Patients With Severe Haemophilia A
Acronym: UK-PK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hampshire Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2015-MED-13
Record Dates: First submitted 2015-07-17; First posted 2015-08-19 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Hemophilia A
Keywords: Pharmacokinetic dosing; Haemophilia
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Educational Package (Other): Patients will receive a standardised PK focused educational package in the form of a short video film.
  Interventions: Behavioral: Educational Package

INTERVENTIONS:
Behavioral: Educational Package — Patients will be invited to attend a PK educational session as part of the study protocol. This will form a discussion regarding clinical history and activity in the 6 months prior to study start, viewing of a short animated film giving additional detail on pharmacokinetics and prophylaxis in haemophilia A, followed by modelling of the patient's own PK and dose guidance based on 2 study blood samples.

SUMMARY:
Prospective, interventional study of pharmacokinetic (PK)-focused FVIII dosing discussions delivered as part of a patient education package.

The study will capture severe haemophilia A patient reported outcome measures before and after PK-focused dosing discussions, including a standardised patient education package, that include personalised PK-guided dosing suggestions from a computational predictive device (myPKFiT®). The pragmatic study design recognises the CE marked myPKFiT® device is being implemented into routine care nationally and consequently only requires a single additional clinic visit for the purpose of consenting.

DETAILED DESCRIPTION:
There is a paucity of patient reported outcome data documenting the impact of PK focused prophylaxis discussions. This prospective, multicentre UK-PK trial will coincide with the initiation of the myPKFiT® device in the context of an enhanced clinical review. This will include a standardised patient education package using a short animated film explaining PK and personalised prophylaxis, followed by modelling of the patient's own PK using the myPKFiT® device and discussing the dosing options with the patient. The aim of the PK educational package is to educate and engage patients and ensure that their treatment regimens meet their individual needs. In addition, the study will capture the prophylaxis dosing strategy agreed upon by patients and the clinical team where treatment decisions are made jointly between patients and the clinical team (concordance). Looking forward, haemophilia clinical care team members need a marker to judge or predict patient engagement with this personalising medicine process. Successful consultation strategies may differ if the team can anticipate how an individual person with haemophilia (PWH) might respond to discussions about potential change. The primary outcome measure is the Patient Activation Measure (PAM) which gauges the knowledge, skills and confidence essential to managing one's own health and healthcare. A PAM score can predict healthcare outcomes including medication adherence, healthcare utilisation and hospital visits. It is hypothesized that a more activated patient will be more receptive to changes in their treatment regimen, education and information about their health condition.

In addition to patient activation, the study will assess a range of patient reported outcomes and psychological factors using validated tools. These will include patients' Haemophilia-related quality of life (HAEMO-QoL-A), beliefs about medicines (BMQ), self-reported adherence (VERITAS-Pro) and activity levels. These tools will provide clear patient reported outcomes for the haemophilia community, with accompanying EQ5D data, enabling robust health economic evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Severe haemophilia A (FVIII:C < 1IU/dL)
* Prescribed regular prophylactic treatment (≥ 2 infusions/week) with Advate® for ≥ 6 months at the time of screening
* Able to give informed consent and willing to participate in this study

Exclusion Criteria:

* Age <18 years
* Non-severe haemophilia A (FVIII:C 1-40IU/dL)
* Weight >120kg
* Treatment with any other FVIII concentrate (recombinant or plasma-derived) during the study period or 6 months prior to screening.
* Receiving on-demand or <6 months of prescribed prophylaxis with Advate®
* Current FVIII inhibitor (> 0.6BU/mL)
* Current immune tolerance induction
* Not able to give informed consent (incapacitated or vulnerable adults)
* Patients with a life expectancy of less than one year
* Already had personalized PK prediction using the myPKFiT®
* Any inclusion criteria not met

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Change in Patient Activation Measures | 12 months
  Change in the Patient Activation Measure (PAM) score over a 12 month time period.

SECONDARY OUTCOMES:
Patients' perceptions of the PK educational package | 12 months
  Perceived threat, message quality, message acceptance/derogation. This will be measured qualitatively.
Health-related quality of life: EQ5D | 12 months
Health-related quality of life: HAEMO-QoL-A | 12 months
Self-reported adherence (VERITAS-pro) | 12 months
Health-related quality of life: beliefs about medicines (BMQ) | 12 months
Changes to participants' treatment regimen | 12 months
  Change to amount of FVIII used
Changes to accuracy and timeliness of entries on treatment log (Haemtrack or alternative treatment log). | 12 months
Changes to patient adherence to treatment regimen | 12 months
  Actual changes as recorded on Haemtrack / equivalent.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Hart, Principal Investigator — Barts & The London NHS Trust
Locations (1):
- Barts and The Royal London Hospital, London, United Kingdom